CLINICAL TRIAL: NCT07355595
Title: The Effect of the Mobile App-Assisted Home Exercise Program on Clinical Outcomes in Patients With Musculoskeletal Disorders
Brief Title: Mobile App-Assisted Home Exercise for Musculoskeletal Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Wendy Tzyy-Jiuan Wang, Professor, Department of Physical Therapy, National Yang Ming Chiao Tung University, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU114207AE
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Disorders; Low Back Pain; Neck Pain; Shoulder Pain; Knee Pain
Keywords: e-Health; Mobile Applications; Home Exercise Program
MeSH Terms: conditions — Musculoskeletal Diseases; Low Back Pain; Neck Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-Assisted Group (Experimental): Participants in this group will receive a 4-week program consisting of weekly physiotherapy sessions and a daily 10-minute home exercise program assisted by a dedicated mHealth application
  Interventions: Behavioral: Mobile App-Assisted Home Exercise with Standard Physiotherapy
- Control Group (Active Comparator): Participants in this group will receive a 4-week program consisting of weekly physiotherapy sessions and a daily 10-minute traditional home exercise program without mobile application support
  Interventions: Behavioral: Traditional Home Exercise with Standard Physiotherapy

INTERVENTIONS:
Behavioral: Mobile App-Assisted Home Exercise with Standard Physiotherapy — Participants will receive one 30-minute face-to-face physiotherapy session weekly for 4 weeks. Concurrently, they will perform a daily 10-minute home exercise program via a dedicated mobile health application that provides automated reminders, home exercise video demonstrations, self-monitoring of exercise data, tele-consultation capabilities, and patient education on pain pathology
  Arms: App-Assisted Group
Behavioral: Traditional Home Exercise with Standard Physiotherapy — Participants will receive one 30-minute face-to-face physiotherapy session weekly for 4 weeks. Concurrently, they will perform a daily 10-minute home exercise program based on verbal instructions provided by the physiotherapist. This group will not have access to any mobile health application or digital support
  Arms: Control Group

SUMMARY:
Overview This study evaluates the effectiveness of a dedicated mobile health (mHealth) application in supporting home exercise programs for patients with musculoskeletal disorders, such as neck, shoulder, back, or knee pain. The research aims to address the widespread challenge of low patient adherence to unsupervised home-based exercises.

Study Design The project employs a dual-methodology approach:

Clinical Trial: 30 participants presenting with neck, shoulder, back, or knee pain will be randomly assigned to either an app-assisted group or a traditional home exercise group. Both groups will undergo 4 weeks of physiotherapy. The study will compare pain intensity, physical function, and exercise adherence between the two cohorts.

Retrospective Analysis: To complement the trial, the study will analyze a large-scale database containing approximately 700,000 anonymized real-world data entries. This analysis aims to observe real-time pain fluctuations before and after exercise sessions within routine clinical settings.

Goal The primary objective is to determine if integrating mHealth technology into traditional rehabilitation can enhance clinical outcomes and improve patient adherence to home-based exercise routines.

DETAILED DESCRIPTION:
Background: Musculoskeletal disorders are a leading cause of disability worldwide. Exercise prescription is a cornerstone of musculoskeletal rehabilitation, and physiotherapists often provide home-based exercise programs as part of self-management strategies. This approach is not only an active adjunctive intervention but also cost-effective. However, according to the 2021 Taiwan National Health Interview Survey, 54% of adults did not meet the World Health Organization's recommended physical activity levels-significantly higher than the global average of 27%-highlighting the low adherence to unsupervised exercise among Taiwanese adults. With the advancement of technology, electronic health (e-Health) interventions have become increasingly prevalent. Smartphone applications can provide reminders, recording, and personalized designs to improve adherence and clinical outcomes. Nonetheless, systematic reviews have reported that most commercially available apps have limited coverage of behavior change intervention functions (BCIFs) and lack rigorous scientific validation, leaving their clinical efficacy and large-scale applicability uncertain. Youdon, a mobile app developed by Meike Tech in Taiwan, aims to enhance accessibility and adherence to home exercise programs among Taiwanese patients. Despite its comprehensive behavior change functions, the app's clinical effectiveness remains to be verified through scientific research.

Purpose: This study aims to investigate the clinical effectiveness of a mobile app-assisted home exercise program in patients with musculoskeletal disorders, through two complementary components:

1. A randomized controlled trial (RCT) comparing pain and functional outcomes between app-assisted and non-assisted home exercise programs.
2. A retrospective observational study analyzing app-user data to evaluate real-time pain changes before and after exercise and their associated factors.

Methods:

Part I: A single-blind randomized controlled trial will recruit 30 participants aged 18 years and above presenting with neck, shoulder, low back, or knee pain. Participants will be randomly assigned to either an app-assisted group or a control group without app support. Both groups will receive a 4-week intervention consisting of weekly physiotherapy sessions and daily 10-minute home exercises. Primary outcomes include pain intensity, Patient-Specific Functional Scale (PSFS) scores, and region-specific disability indices; the secondary outcome is exercise adherence. Measurements will be conducted at baseline, week 2, and week 4. Data will be analyzed using an intention-to-treat approach and mixed ANOVA to examine time and group effects (p < 0.05).

Part II: A retrospective observational study will analyze approximately 700,000 anonymized data entries from the Youdon database between July 1, 2024, and August 30, 2025. The study will assess real-time changes in pain before and after each exercise session and identify influencing factors under routine clinical conditions. Data will be analyzed using linear mixed-effects models (LMMs), with participant ID set as a random intercept to account for within-subject variability.

Model 1 (Pain improvement model): The dependent variable will be the pain change score; predictors include functional diagnosis, number of pain sites, pre-exercise pain score, and exercise adherence.

Model 2 (Adherence model): The dependent variable will be exercise adherence; predictors include number of pain sites, pre-exercise pain, number of exercise prescriptions, and perceived exertion. Both models will adjust for age and sex as covariates.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* Presenting with musculoskeletal disorders leading to pain in the neck, shoulder, low back, or knee
* Scoring 3 or higher on the Numeric Pain Rating Scale

Exclusion Criteria:

* Diagnosis of malignant tumors
* Presence of serious systemic or neurological conditions that may interfere with assessment or treatment, such as uncontrolled hypertension, serious cardiac diseases, or Parkinson's disease
* Inability to use a mobile smartphone
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline, Week 2, and Week 4
  Measured using the Numeric Rating Scale, where scores range from 0 (no pain) to 10 (worst possible pain)
Functional performance | Baseline, Week 2, and Week 4
  Measured using the Patient-Specific Functional Scale (PSFS). Participants identify at least three activities that are most affected by their condition and rate their ability to perform each on an 11-point scale ranging from 0 to 10 (0 = unable to perform activity, 10 = able to perform activity without any difficulty). Higher scores indicate a better functional outcome.
Neck Disability (Neck Disability Index, NDI) | Baseline, Week 2, and Week 4
  Neck-related disability will be assessed using the Neck Disability Index (NDI). The NDI consists of 10 items, each scored on a 6-point scale ranging from 0 to 5, yielding a total score from 0 to 50. The total score will be converted to a percentage score (0-100%), with higher scores indicating a greater degree of functional disability.
Low Back Disability (Oswestry Disability Index, ODI) | Baseline, Week 2, and Week 4
  Low back-related disability will be assessed using the Oswestry Disability Index (ODI). The ODI consists of 10 items, each scored from 0 to 5, resulting in a total score ranging from 0 to 50. The total score will be converted to a percentage score (0-100%), with higher scores indicating a greater degree of functional disability.
Shoulder Disability (Shoulder Pain and Disability Index, SPADI) | Baseline, Week 2, and Week 4
  Shoulder-related disability will be assessed using the Shoulder Pain and Disability Index (SPADI). The SPADI consists of 13 items, including 5 pain items and 8 disability items, each rated on an 11-point numeric rating scale (0-10). Item scores are summed to yield a total score ranging from 0 to 130, which is converted to a percentage score (0-100%) by dividing the total score by 130 and multiplying by 100. Higher scores indicate a greater degree of functional disability.
Knee Disability (International Knee Documentation Committee Subjective Knee Evaluation Form, IKDC) | Baseline, Week 2, and Week 4
  Knee-related disability will be assessed using the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form. The IKDC consists of 18 items covering symptoms, sports activities, and function, of which item 10a is excluded from scoring, yielding a raw score ranging from 0 to 87. The raw score is converted to a standardized score (0-100) by dividing the total score by 87 and multiplying by 100, with higher standardized scores indicating better knee function. For analytical purposes, the standardized IKDC score will be reversed (100 - score), such that higher transformed scores indicate a greater degree of functional disability.

SECONDARY OUTCOMES:
Exercise Adherence | Daily for 4 weeks
  Exercise adherence is evaluated using a standardized electronic self-report record form. All participants are required to record real-time data after each home exercise session, including the actual duration of exercise performed (excluding rest periods), pain intensity before and after exercise, and perceived exertion levels. Adherence is defined as the percentage of the actual exercise duration relative to the prescribed duration. A higher percentage reflects better adherence to the home exercise program.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data. The decision may be re-evaluated upon study completion or at the time of publication